CLINICAL TRIAL: NCT04311294
Title: Development of a Selective ALDH2 Inhibitor for the Treatment of Alcohol Use Disorder
Brief Title: Development of a Selective ALDH2 Inhibitor to Treat AUD
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Project was not funded.
Sponsor: University of California, Los Angeles (Other)
Collaborators: Amygdala Neurosciences (Unknown); National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Lara Ray, PhD, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1R21AA028444
Record Dates: First submitted 2020-03-11; First posted 2020-03-17 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Medications Development
MeSH Terms: conditions — Alcoholism | interventions — ANS-6637

STUDY DESIGN:
Intervention Model Description: Randomized, triple-blind, placebo-controlled, parallel-group study of ANS-6637 (200mg, 600mg, 0mg [palcebo])
Who Masked: Participant, Care Provider, Investigator
Masking Description: The study team, medical personnel, and participants will be blind to drug condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ANS-6637 Low Dose (Active Comparator): 200mg ANS-6637 (2 tablets)
  Interventions: Drug: ANS-6637 Low Dose
- ANS-6637 High Dose (Active Comparator): 600mg ANS-6637 (2 tablets)
  Interventions: Drug: ANS-6637 High Dose
- Placebo (Placebo Comparator): 0mg matched placebo (2 tablets)
  Interventions: Drug: Matched Placebo

INTERVENTIONS:
Drug: ANS-6637 Low Dose — ANS-6647 is a selective, reversible, and orally bioavailable aldehyde dehydrogenase 2 (ALDH2) inhibitor. It will be tested at a low dose (200mg) and a high dose (600mg) against matched placebo.
  Arms: ANS-6637 Low Dose
Drug: ANS-6637 High Dose — ANS-6647 is a selective, reversible, and orally bioavailable aldehyde dehydrogenase 2 (ALDH2) inhibitor. It will be tested at a low dose (200mg) and a high dose (600mg) against matched placebo.
  Arms: ANS-6637 High Dose
Drug: Matched Placebo — ANS-6647 is a selective, reversible, and orally bioavailable aldehyde dehydrogenase 2 (ALDH2) inhibitor. It will be tested at a low dose (200mg) and a high dose (600mg) against matched placebo.
  Arms: Placebo

SUMMARY:
Alcohol use disorder (AUD) represents a highly prevalent, costly, and often untreated condition in the United States. Pharmacotherapy offers a promising avenue for treating AUD and for improving clinical outcomes for this debilitating disorder. While developing novel medications to treat AUD remains a high priority research area, there are major opportunities to refine the process of screening novel compounds.

A promising novel pharmacology for AUD consists of the ANS-6637 compound which provides novel aldehyde dehydrogenase 2 (ALDH2) inhibition. Unlike disulfiram, a non-selective and irreversible ALDH2 and ALDH1 inhibitor, which produces an aversive flushing response, the oral ANS-6637 compound is a selective and reversible inhibitor of ALDH2 that attenuates the surge in dopamine (DA). Specifically, a preclinical study found that ANS-6637 blunted the surge of DA in ventral tegmental neurons without affecting the basal levels of DA in vivo in a rodent model of alcohol seeking behavior. In rodent models, selective and reversible ALDH2 inhibitors decrease alcohol seeking and taking, prevent operant self-administration, and block cue-induced reinstatement. These results suggest that ANS-6637 may be an effective treatment to reduce heavy drinking and suppress relapse in individuals with AUD.

This is a randomized, double-blind, placebo-controlled, dose response study of ANS-6637. A total of 75 men and women with current AUD will be randomly assigned to receive (a) ANS-6637 (200 mg), (b) ANS-6637 (600 mg), or (c) matched placebo for 7 days. On Day 4, participants will complete an fMRI task before and 45-minutes after a priming dose of alcohol (target Breath Alcohol Concentration (BrAC) of 0.03 g/dl). On Day 7 participants will return to the laboratory to complete an oral alcohol administration paradigm. The successful completion of this study will advance medications development for AUD by advancing the development of ANS-6637, a novel and promising compound for AUD.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years and older (adult, older adult);
2. meeet DSM-5 diagnostic criteria for alcohol use disorder (moderate or severe);
3. report drinking at least 48 standard drinks in a 30-day period, during the 90 days before enrollment.

Exclusion Criteria:

1. current treatment for alcohol problems;
2. a history of treatment for alcohol problems in the 30 days before enrollment;
3. currently seeking treatment for alcohol problems;
4. current DSM-5 diagnosis of dependence on any psychoactive substances other than alcohol or nicotine;
5. lifetime DSM-5 diagnosis of schizophrenia, bipolar disorder, or any psychotic disorder;
6. positive urine screen for narcotics, amphetamines, or sedative hypnotics;
7. serious alcohol withdrawal symptoms as indicated by a score of ≥10 on the Clinical Institute Withdrawal Assessment for Alcohol-Revised (CIWA-Ar)
8. pregnant, nursing, or refusal to use reliable birth control method (if female);
9. medical condition that may interfere with safe study participation (e.g. unstable cardiac, renal, or liver disease, uncontrolled hypertension or diabetes);
10. AST, ALT, or GGT ≥ 3 times upper limit of normal;
11. attempted suicide in the past 3 years and/or serious suicidal intention or plan in the past year;
12. currently on prescription medication that contraindicates use of ANS-6637;
13. other circumstances that, in the opinion of the investigators, compromises participant safety

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-04 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Change in Subjective Response to Alcohol | Baseline, 30-, 45-, 60-, 120-, and 180-minutes post alcohol
  Participants will complete an oral alcohol challenge and will rate their subjective responses to alcohol at baseline (BrAC = 0.00 g/dl) and at 30, 45, 60, 120, and 180 minutes post alcohol. The primary outcome variables will be (a) alcohol craving, (b) stimulant/reward, and (c) sedative/aversive effects of alcohol.
Change in Neural Alcohol Cue Reactivity | Assessed on Day 4. Scan duration 1 hour.
  Participants will complete a neuroimaging paradigm in which they view alcoholic and non-alcoholic beverage cues and will rate their subjective craving for alcohol. The primary outcome variable will be BOLD activation to alcohol cues in mesocorticolimbic reward circuitry.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Ray, PhD, Principal Investigator — University of California, Los Angeles; Erica Grodin, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Addictions Lab, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
All data collected in this project will be shared (after appropriate de-identification) with the scientific community in a timely manner, in accordance with NIH Policy. Specifically, the dataset will be made available to the scientific community upon request and a data application will be required. These procedures are consistent with the recent NIAAA announcement: NOT-AA-18-010